CLINICAL TRIAL: NCT00534547
Title: Phase IV Study of Duodenal Exclusion for the Treatment of Type 2 Diabetes (T2DM)
Brief Title: Duodenal Exclusion for the Treatment of Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: business reasons
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS07009
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Duodenal Exclusion — duodenal-jejunal bypass

SUMMARY:
The purpose of this study is to investigate the role of an experimental surgery that may offer better short and long-term control of T2DM in select patients who have not achieved adequate blood sugar control with regular means.

ELIGIBILITY:
Inclusion criteria:

* Age between 20 and 50 years old;
* BMI between 27 and 34.9;
* Oral agents or insulin to control T2DM;
* Inadequate control of diabetes as defined as HbA1c>8.0% but <10%
* Understanding of the mechanisms of action of the treatment

Exclusion criteria:

* More than 5 years of T2DM diagnosis;
* C-peptide <1pg/ml (off insulin)
* Previous abdominal operations;
* History of gastritis
* History of GERD
* History of peptic ulcer disease
* Inflammatory bowel disease
* Coagulopathy;
* Liver cirrhosis;
* Unable to comply with study requirements, follow-up schedule or give valid informed consent;
* Currently pregnant (pregnancy test required for confirmation for those of child bearing years)
* Patient is not available for programmed follow-up during the study period
* Patient is unwilling to forgo good samaritan blood donation during the study period

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Treatment success based on patients' glycemic control | 12 Months

SECONDARY OUTCOMES:
Physiologic Measurements, Comorbidity improvement, Improvement in QOL | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Fahey, Study Director — Medtronic - MITG